CLINICAL TRIAL: NCT06180148
Title: Use of Mechanical Insufflator-exsufflator in Patients After Video-assisted Thoracoscopic Operations With One-lung Ventilation on Postoperative Pulmonary Complications: a Randomized Trial
Brief Title: Mechanical Insufflator-exsufflator in Patients After Video-assisted Thoracoscopic Operations With One-lung Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COUGH-001
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2023-12

CONDITIONS: Thoracic Diseases
Keywords: One-lung ventilation; Postoperative pulmonary complications; Mechanical insufflator-exsufflator; Randomized trial
MeSH Terms: conditions — Thoracic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mechanical insufflator-exsufflator (Active Comparator): Standard postoperative care plus mechanical insufflator-exsufflator during the first postoperative day.
  Interventions: Device: Mechanical insufflator-exsufflator
- Standard care (No Intervention): Standard postoperative care without mechanical insufflator-exsufflator.

INTERVENTIONS:
Device: Mechanical insufflator-exsufflator — In the active comparator group a mechanical insufflator-exsufflator will be used in the postoperative period 6 and 24 hours after extubation as follows ("coughing maneuver"): application of inspiratory pressure of 40-70 cm of water (the minimum value to achieve a peak cough flow of 300 l/min) for 2 seconds with the subsequent creation of an expiratory vacuum of -40 cm of water within 2 seconds. During inhalation and exhalation, the patient will apply oscillations with a frequency of 10 Hz and an amplitude of 10 cm of water. A series of 10 such maneuvers will be used, with a pause of a few seconds to ensure patient comfort. The "coughing" maneuver will be performed through an oronasal mask tightly pressed to the face.
  Arms: Mechanical insufflator-exsufflator

SUMMARY:
Postoperative pulmonary complications (PPC) are a common problem in patients undergoing surgery using one-lung invasive ventilation. Major pulmonary complications such as atelectasis, bronchospasm, and pneumonia can lead to respiratory failure. PPC are the main cause of mortality in the postoperative period in patients after thoracic surgery. The study aimed to compare the effectiveness of using a mechanical insufflator-exsufflator after video-assisted thoracoscopic surgery using one-lung ventilation to reduce postoperative pulmonary complications as compared to standard therapy.

DETAILED DESCRIPTION:
Postoperative pulmonary complications (PPC) are a common problem in patients undergoing surgery using one-lung invasive ventilation. Major pulmonary complications such as atelectasis, bronchospasm, and pneumonia can lead to respiratory failure. PPC are the main cause of mortality in the postoperative period in patients after thoracic surgery. The incidence of PPC ranges from 5% to 80%. Patients undergoing thoracic surgery are usually at high risk. Most often these are elderly people with concomitant diseases. Most of these patients are smokers, have occupational exposures, and are therefore at even greater risk of developing pulmonary complications. Part of their problem is due to poor baseline pulmonary function. Improving mucus production in the postoperative period using a mechanical insufflator-exsufflator may help reduce the incidence of complications.

ELIGIBILITY:
Inclusion Criteria:

* Video-assisted thoracoscopic surgery using one-lung ventilation
* Age 18-65 years Forced expiratory volume in one second (FEV1) 60% of predicted or more
* Absence of pronounced bronchial secretion before surgery
* Written informed consent.

Exclusion Criteria:

* Age less than 18 and more than 65 years
* Presence of pneumothorax 6 hours after surgery on radiography
* Pulmonary hemorrhage of any intensity
* Unstable hemodynamics
* Forced expiratory volume in one second (FEV1) is less than 60% of predicted during preoperative examination
* The scope of the operation is more than a lobectomy
* Bilateral and combined operations
* Mechanical ventilation after surgery for more than 6 hours
* Anesthesia risk according to American Society of Anesthesiologists (ASA) 4 and 5 points

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2024-01-09 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Peripheral oxygen saturation level (SpO2) when breathing atmospheric air 6 hours after tracheal extubation | On 6 hour after operation
  Peripheral oxygen saturation level (SpO2) when breathing atmospheric air 6 hours after tracheal extubation
Peripheral oxygen saturation level (SpO2) when breathing atmospheric air 24 hours after tracheal extubation | On 24 hour after operation
  Peripheral oxygen saturation level (SpO2) when breathing atmospheric air 24 hours after tracheal extubation
Sputum volume 24 hours after tracheal extubation | On 24 hour after operation
  Sputum volume 24 hours after tracheal extubation
Peak expiratory flow (PEF) 48 hours after surgery | On 48 hour after operation
  Peak expiratory flow (PEF) 48 hours after surgery,
The volume of atelectasis on chest computed tomography 36-48 hours after tracheal extubation | On 36-48 hour after operation
  The volume of atelectasis on chest computed tomography 36-48 hours after tracheal extubation

SECONDARY OUTCOMES:
Pain according to visual analogue scale (VAS) of pain 6 hours after tracheal extubation | On 6 hour after operation
  Pain according to visual analogue scale (VAS) of pain 6 hours after tracheal extubation (from 1 to 10 points, where 1 point - minimal pain level, 10 points - maximal pain level)
Pain according to visual analogue scale (VAS) of pain 24 hours after tracheal extubation | On 24 hour after operation
  Pain according to visual analogue scale (VAS) of pain 24 hours after tracheal extubation (from 1 to 10 points, where 1 point - minimal pain level, 10 points - maximal pain level)
Dyspnea according to visual analogue scale (VAS) of dyspnea 6 hours after tracheal extubation | On 6 hour after operation
  Dyspnea according to visual analogue scale (VAS) of dyspnea 6 hours after tracheal extubation (from 1 to 10 points, where 1 point - minimal comfort, 10 points - maximal comfort)
Dyspnea according to visual analogue scale (VAS) of dyspnea 24 hours after tracheal extubation | On 24 hour after operation
  Dyspnea according to visual analogue scale (VAS) of dyspnea 24 hours after tracheal extubation (from 1 to 10 points, where 1 point - minimal comfort, 10 points - maximal comfort)
Postoperative pulmonary complications | Day 7 after operation
  Development of postoperative pulmonary complications - atelectasis (focus of consolidation on CT scan of the lungs without signs of infection), respiratory tract infection - tracheobronchitis or pneumonia (CPIS score>5 points), hypoxemia (SpO2<90% when breathing atmospheric air), pleural effusion (more than 300 ml), pneumothorax, bronchospasm (clinically - the presence of dry wheezing).

CONTACTS AND LOCATIONS:
Locations (1):
- Sechenov University Clinic#4, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No